CLINICAL TRIAL: NCT01921868
Title: An Open-label Study of the Effects of Acetyl-L-Carnitine on Cardiovascular Outcomes in Friedreich's Ataxia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Theresa Zesiewicz, Professor, Director of USF Ataxia Research Center, University of South Florida
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALCAR-8499
Record Dates: First submitted 2013-07-03; First posted 2013-08-13 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Friedreich's Ataxia
MeSH Terms: conditions — Friedreich Ataxia | interventions — Acetylcarnitine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acetyl-L-Carnitine (Experimental): Open-label administration of Acetyl-L-Carnitine, up to 2 g/day for 24 months.
  Interventions: Drug: Acetyl-L-Carnitine

INTERVENTIONS:
Drug: Acetyl-L-Carnitine — Acetyl-L-Carnitine, 2 g/day, up to 24 months.
  Other Names: ALCAR

SUMMARY:
The purpose of this study is to learn how treatment with acetyl-L-carnitine (ALCAR) will affect the hearts of patients with Friedreich's Ataxia as well as how it may affect other symptoms of Friedreich's Ataxia such as difficulties with balance, walking, or upper arm function.

DETAILED DESCRIPTION:
This study is an open label, pilot study of ALCAR in subjects with FA. In this study 20 patients with FA will receive ALCAR every day for 24 months. At the study endpoint, subjects will be assessed for changes in cardiovascular outcomes and FA symptoms. To determine the effects of LC on changes in cardiomyopathy, echocardiography with strain rate will be calculated. This technique has been validated in clinical studies and used in other studies of FA patients for the comparison of regional deformation and myocardial wall thickness.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients with Friedreich's Ataxia diagnosed by a movement disorder specialist and confirmed by genetic testing (of the patient or in a first degree relative of the patient). Subject may be non-ambulatory.
2. Age 18 years to 80 years.
3. Stable medical condition for 3 months prior to screening.
4. Women of child-bearing potential must use a reliable method of contraception and must provide a negative pregnancy test at entry into the study.
5. If on cardiac medications such as beta-blockers or ace inhibitors, patients must be on a stable dose for 6 months prior to study entry and for the duration of the study.
6. Friedreich's Ataxia patients with systolic or diastolic dysfunction present on echocardiogram and ejection fraction between 35% - 65% at screening.
7. Subjects with ejection fractions < 50% need to be stable and on optimal heart failure therapy for at least 2 weeks prior to screening.

Exclusion Criteria:

1. Any unstable illness or concomitant medical condition that, in the investigator's opinion, precludes participation in this study. This includes other disorders that may affect gait or balance (stroke, arthritis, etc).
2. Pregnancy or lactation.
3. Concurrent participation in another clinical study where use of an investigational product is used. Subjects who are currently enrolled in the Friedreich's Ataxia Clinical Outcome Measures Study at any site will be allowed to enroll in this study as well.
4. Any use of the investigational product within the past 30 days.
5. Dementia or other psychiatric illness that prevents the patient from giving informed consent (Mini Mental Status Exam score less than 25).
6. Legal incapacity or limited legal capacity.
7. History of stroke.
8. Subjects with a history of thyroid disease (hypothyroidism). Clinical laboratory evaluations of thyroid stimulating hormone levels taken 3 months prior to the study or at screening will be used to confirm absence of current thyroid problems.
9. Subjects with a history of seizures.
10. Subjects taking warfarin or acenocoumarol.
11. Presence of severe renal disease (estimated creatinine clearance <50 mL/min) or hepatic disease (AST or Alanine transaminase(ALT)>2x times normal) (as evidenced by labs reported within the past 6 months).
12. Clinically significantly abnormal white blood cell, hemoglobin or platelet count (as evidenced by labs reported within the past 6 months).
13. Subjects with blood work showing carnitine deficiency (<60nmol/mg total carnitine in the urine or <35umol/L total carnitine in the plasma).

    -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-08; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
To observe the changes in cardiac functioning in patients with Friedreich's Ataxia between study endpoint and baseline. | Every 12 months, up to 24 months
To assess the changes in Friedreich's Ataxia symptoms and severity (as measured by clinical rating scales) compared to baseline. | Every 6 months, up to 24 months

SECONDARY OUTCOMES:
Changes in patient global impression of improvement | Every 6 months, up to 24 months
Changes in Time 25-foot Walk | Every 6 months, up to 24 months
Changes in frequency and severity of adverse events | Every 6 months, up to 24 months
Changes in patient quality of life (SF-36) | Every 6 months, up to 24 months
Changes in clinical global impression of improvement | Every 6 months, up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Theresa A Zesiewicz, MD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States